CLINICAL TRIAL: NCT04494451
Title: Efficacy of Vitamin C on AKI Outcomes in Critically Ill Cirrhotics With Multidrug-resistant Bacterial Infections- A Randomized Controlled Trial
Brief Title: Efficacy of Vitamin C on AKI Outcomes in Critically Ill Cirrhotics With Multidrug-resistant Bacterial Infections.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis-35
Record Dates: First submitted 2020-07-28; First posted 2020-07-31 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-10

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin C + Standard Medical Treatment (Experimental): vitamin C (25 mg/kg or max. 1.5 gram every 6 hourly) for maximum 5 days along with iv antibiotics as per institutional protocol along with iv antibiotics
  Interventions: Drug: Vit C; Drug: Standard medical Treatment
- Standard Medical Treatment (Active Comparator): iv antibiotics alone
  Interventions: Drug: Standard medical Treatment

INTERVENTIONS:
Drug: Vit C — vitamin C (25 mg/kg or max. 1.5 gram every 6 hourly) for maximum 5 day
  Arms: Vitamin C + Standard Medical Treatment
Drug: Standard medical Treatment — iv antibiotics alone

SUMMARY:
In this prospective randomized controlled trial we aim to evaluate the impact of vitamin C on AKI outcomes in patients with cirrhosis and MDR infections. We also aim to evaluate the effects of iv vitamin c on systemic hemodynamics (cardiac output and systemic vascular resistive index, extravascular lung water and lung permeability index), endothelial function and coagulation, microcirculation (as assessed by lactate clearance and central venous oxygen saturation), mitochondrial function, 28-day mortality and vasopressor, ventilator and RRT free days in the ICU. The safety and side-effects of vitamin c would also be evaluated.

Patients with suspected (nosocomial acquisition) or proven MDR infections would be screened and randomized to two groups who meet the inclusion and exclusion criteria.

Group 1: Will receive iv vitamin C (25 mg/kg or max. 1.5 gram every 6 hourly) for maximum 5 days along with iv antibiotics as per institutional protocol Group 2: iv antibiotics alone

DETAILED DESCRIPTION:
Aim & Objectives Primary To evaluate the impact of vitamin C on AKI outcomes in patients with cirrhosis and MDR infections

Secondary Objectives To assess the effects on systemic hemodynamics (cardiac output and systemic vascular resistive index, extravascular lung water and lung permeability index) Impact of Vitamin C on endothelial function and coagulation Improvement in microcirculation as assessed by lactate clearance and central venous oxygen saturation To assess the effects on 28-day mortality. Improvement in SOFA scores in both groups Vasopressor, ventilator and RRT free days in the ICU Incidence of adverse effects in both groups Prevalence of vitamin C deficiency in cirrhotics with sepsis and impact of exogenous vitamin C in improving endogenous levels of ascorbate and norepinephrine levels Impact of vitamin C on oxidative stress by evaluation of mitochondrial bioenergetics

(B) Methodology Patients with suspected (nosocomial acquisition) or proven MDR infections would be screened and randomized to two groups as under Group 1: Will receive iv vitamin C (25 mg/kg or max. 1.5 gram every 6 hourly) for maximum 5 days along with iv antibiotics as per institutional protocol Group 2: iv antibiotics alone All patients with nosocomial bacterial infections or septic shock would be screened for randomization would be considered for enrolment in the trial. Nosocomial infection would be defined as infections developing after 48 hours of hospitalization. Following this, patients meeting the inclusion and exclusion criteria will be screened and randomized to the two treatment groups. Standard of care for management of antibiotics, fluids and vasopressors would be as per institutional guidelines. At baseline, blood and urine sample would be stored for all patients for performing mitochondrial bioenergetics, endotoxin, proinflammatory cytokines (IL-6, IL-IB, TNF-alpha, MCP-1, IL-1O) and urine biomarkers (urine NGAL and cystatin C) and markers of endothelial dysfunction(von willebrand factor and ADAMTS). Following randomization patients would be allocated to receive intravenous vitamin C (1.5 g every 6 h or 25 mg/kg for 5 days) along with intravenous antibiotics

Study Population:

Patients with cirrhosis with MDR infections (nosocomial acquisition) or culture-proven

Study Design:

* A randomized controlled study.
* The study will be conducted on patients admitted to Department of Hepatology from June 2020 to December 2020 at ILBS, New Delhi
* Study group will comprise of patients critically ill cirrhotics with suspected or proven MDR infections

Study period

* The study will be conducted on patients admitted to Department of Hepatology from June 2020 to December 2020 at ILBS, New Delhi
* Study group will comprise of patients critically ill cirrhotics with MDR infections.

Sample Size calculation: Currently there are lack of studies investigating the incidence and outcomes of AKI in this context. The study will be designed as a pilot RCT with an aim to enrol 50 patients in each group.

The detailed cytokine profile, endotoxin assay, markers of endothelial dysfunction and bioenergetics would be performed in a subset of 15 patients in each group.

Intervention: IV Vitamin C

Monitoring and Assessment: Hourly till the patient is in the intensive care unit then every 7 days for 1 month

Statistical analysis

* All variables shall be expressed in mean (sd) or median (range)
* Variables will be compared by Mann- Whitney U test
* For Categorical variables we will use Chi-Square or Fisher's test
* Survival analysis will be done using Cox-proportional regression analysis

Actuarial probability of survival shall be calculated by Kaplan- Meier graph and compared by log- rank test.

Adverse Effects: Any allergic reactions, drop in hemoglobin or development of kidney stones

Stopping rule of the study: Any untoward adverse effects of the intervention.

Ethical issues in the study and plans to address these issue The study is designed to demonstrate the efficacy of intravenous vitamin C in improving AKI outcomes in cirrhotics with MDR infections. Vitamin C is been routinely used in this indication with no major adverse effects. However, head-to-head comparison is needed to identify the evidence and benefits of using this drug in this indication. Only minor side effects like nausea, diarrhea, abdominal bloating, cramps and precipitation of kidney stones have been observed with the drug.

ELIGIBILITY:
Inclusion Criteria:

- Critically ill cirrhotics with MDR infections

Exclusion Criteria:

* Patients with age less than 18 years
* Known severe cardiopulmonary disease (structural or valvular heart disease, coronary artery disease, COPD)
* Patients in DIC with platelets < 20,000 and INR > 4 or active bleeding
* Limitations of care (defined as refusal of cardiovascular and respiratory support modes) including "do not intubate" (DNI) status
* Current hospitalization > 15 days for patients with nosocomial acquisition of MDR at time of randomization
* Known allergy or contraindication to vitamin C (including previously or currently diagnosed primary hyperoxaluria and/or oxalate nephropathy, or known/suspected ethylene glycol ingestion,
* Known glucose-6-phosphate dehydrogenase (G6PD) deficiency)
* Use of vitamin C at a dose of > 1 gram daily within the 24 hours preceding first episode of qualifying organ dysfunction during a given ED or ICU admission
* Patients with HCC (beyond Milan) or extrahepatic malignancies
* Patients with HVOTO or EHPVO
* Pregnancy or active breastfeeding
* Current participation in another interventional research study
* Active or history of kidney stone
* History of chronic kidney disease or intrinsic kidney disease
* Patients already on maintenance hemodialysis prior to presentation
* Patients with refractory septic shock or hypoxemia (Pa02/Fio2 ratio <100)
* Extremely moribund patients with an expected life expectancy of less than 24 hours
* Failure to provide informed consent
* Patients with retroviral infection
* Patients with acute on chronic liver failure (APASL definition)
* Patients with urinary tract infection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-11-02 (Actual); Study Completion 2022-11-02 (Actual)

PRIMARY OUTCOMES:
AKI progression at day 5 | Day 5

SECONDARY OUTCOMES:
Mortality in both groups | Day 28
Time to reversal of AKI in both groups | Day 14
Lactate clearance in both groups | 12 hours
Lactate clearance in both groups | 24 hours
Vasopressor, ventilator and days free of dialysis during ICU stay | Day 28

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided